CLINICAL TRIAL: NCT00107601
Title: A Multi-Center Study Comparing the Effects of Two Glucose Control Regimens by Insulin in Intensive Care Unit Patients
Brief Title: Glucontrol Study: Comparing the Effects of Two Glucose Control Regimens by Insulin in Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Belgian Government (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-003914-40; EUDRACT Number: 200400391440
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2006-02

CONDITIONS: Critical Illness
Keywords: Glucose; Glucose Control; Insulin; Insulin therapy; Critically ill; Intensive Care
MeSH Terms: conditions — Critical Illness; Insulin Resistance | interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
Glucontrol is a prospective, randomized, controlled, multi-centric study. The present study will compare the effects of two regimens of insulin therapy, respectively titrated to achieve a blood sugar level between 4.4 and 6.1 mmol/l (80 and 110 mg/dl, respectively) and between 7.8 and 10.0 mmol/l (140 and 180 mg/dl, respectively).

This project aims at defining whether a tight glucose control by insulin improves the vital outcome in a mixed population of critically ill patients (around 3000 patients).

Secondary outcome variables will include in-hospital and 28-day mortality, lengths of stays in the Intensive Care Unit (ICU) and in the hospital, length of ICU stay without life-support therapy, number and clinical signs of episodes of hypoglycemia, rates of infections and organ failures, and number of red-cell transfusions.

DETAILED DESCRIPTION:
Hyperglycemia frequently occurs during critical illness and is commonly implicated in the development of potentially lethal infectious, vascular and metabolic complications. We hypothesize that a control of glycemia by insulin will improve the vital outcome and the rate of complications in a heterogeneous population of critically ill patients. This hypothesis is supported by the findings of a recent trial performed in one surgical intensive care unit, which demonstrated a significant improvement in vital outcome and in several indices of morbidity in patients randomized to a tight control of glycemia. However, these findings can hardly be extrapolated to other conditions, including different types of pathologies and management. The present prospective, randomized, controlled and multicentric study, will compare the effects of two regimens of insulin therapy, respectively titrated to achieve a blood sugar level between 4.4 and 6.1 mmol/l (80 and 110 mg/dl, respectively) and between 7.8 and 10.0 mmol/l (140 and 180 mg/dl, respectively) and will be powered to detect a 4% decrease in absolute intensive care unit (ICU) mortality. Secondary outcome variables will include in-hospital and 28-day mortality, lengths of stays in ICU and in the hospital, length of ICU stay without life-support therapy, number and clinical signs of episodes of hypoglycemia, rates of infections and organ failures, number of red-cell transfusions.

ELIGIBILITY:
Inclusion Criteria:

* All adult (older than 18 years old at admission) patients admitted in Intensive Care Unit whatever the reason

Exclusion Criteria:

* Absence of the informed consent (as approved by the local ethical committee).
* Life expectancy lower than 24 hours, as estimated upon admission.
* Therapeutic limitation upon admission in ICU
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500
Dates: Start 2004-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Mortality in the Intensive Care Unit (ICU)

SECONDARY OUTCOMES:
Hospital mortality
28 Day mortality
Length of ICU stay
Length of hospital stay
Number of episodes of hypoglycemia and associated clinical signs
Infectious morbidity
Incidence of organ failures
Number of red-cell transfusions
Number of days spent in ICU without life-support: vasopressors/inotropes, cardiac mechanical support, mechanical ventilation, renal replacement therapy
Daily SOFA (Sequential Organ Failure Assessment) Score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devos, Principal Investigator — University of Liege
Locations (11):
- Belgium (3):
  - C.H.U. Erasme, Brussels
  - University Hospital Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- France (3):
  - Hopital Raymond Poincare, Garches
  - Université Joseph Fournier, Grenoble
  - Institut Gustave Roussy, Villejuif
- Universität Ulm, Ulm, Germany
- Rabin Medical Center, Patah Tiqwa, Israel
- V.U.Z. Amsterdam, Amsterdam, Netherlands
- Hospital Universitario General Negrin, Las Palmas de Gran Canaria, Spain
- C.H.U. Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Crosara IC, Melot C, Preiser JC. A J-shaped relationship between caloric intake and survival in critically ill patients. Ann Intensive Care. 2015 Dec;5(1):37. doi: 10.1186/s13613-015-0079-3. Epub 2015 Nov 5. PMID 26541344
- [Derived] Preiser JC, Devos P, Ruiz-Santana S, Melot C, Annane D, Groeneveld J, Iapichino G, Leverve X, Nitenberg G, Singer P, Wernerman J, Joannidis M, Stecher A, Chiolero R. A prospective randomised multi-centre controlled trial on tight glucose control by intensive insulin therapy in adult intensive care units: the Glucontrol study. Intensive Care Med. 2009 Oct;35(10):1738-48. doi: 10.1007/s00134-009-1585-2. Epub 2009 Jul 28. PMID 19636533